CLINICAL TRIAL: NCT00779636
Title: Efficacy and Safety of Desloratadine 10 mg Daily vs. Placebo in Subjects With Allergic Airway Disease During the Pollen Season
Brief Title: Effectiveness and Safety of Desloratadine in Patients With Allergic Airway Disease During the Pollen Season (Study P03284)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03284
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Allergic Airway Disease
MeSH Terms: interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desloratadine 10 mg (Experimental)
  Interventions: Drug: Desloratadine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desloratadine — Desloratadine 10 mg daily x 28 days
  Other Names: Clarinex, SCH 034117
  Arms: Desloratadine 10 mg
Drug: Placebo — Placebo daily x 28 days
  Arms: Placebo

SUMMARY:
This was a placebo controlled study designed to evaluate the effectiveness of desloratadine in relieving symptoms of allergic airway disease during the pollen season. Patients received desloratadine 10 mg or placebo once daily for 28 days, and had their allergy symptoms and side effects to medication measured on Day 1, Day 15, and Day 29 (one day after stopping study drug).

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old
* at least a two-year history of seasonal allergic rhinitis and the presence of chest symptoms (cough, wheezing, difficulty breathing) associated with the allergy season
* FEV1 was greater than or equal to 70% of predicted
* skin test positive (skin prick test)
* Total Nasal Symptom Severity Score of >= 6 at the Screening Visit.
* Total Chest Symptom Severity Score of >= 3 at the Screening Visit.
* Total Frequency of Chest Symptoms and/or Total Frequency of Bronchodilator Use of at least 2 at the Screening Visit
* Total Nasal Symptom Severity Score was >= 6 on 7 of the 15 run-in diary timepoints.
* Total Chest Symptom Severity Score was >= 3 on 7 of the 15 run-in diary timepoints
* Free of any clinically significant disease that would interfere with the study evaluations.

Exclusion Criteria:

Subjects who:

* demonstrated a change in FEV1 of >= 20% between Visit 2 and Visit 3.
* used >12 puffs of Proventil® HFA (or other beta-2-agonist) on any 2 consecutive days or treatment with nebulized beta-2 agonists during the screening period - between Visit 2 and Visit 3.
* required chronic use of inhaled or systemic corticosteroids.
* required regular treatment with nebulized beta2-agonists.
* required short acting beta-2 agonists use before every exercise session or exposure to an animal.
* have current or history of frequent (2 or more episodes per year for the past 2 years), clinically significant sinusitis or chronic purulent postnasal drip.
* have rhinitis medicamentosa or chronic obstructive pulmonary disease (COPD).
* had an upper or lower respiratory tract or sinus infection that required antibiotic therapy with the last dose 14 days prior to Screening, or who have had a upper or lower viral respiratory infection within 7 days prior to Screening.
* had nasal structural abnormalities, including large nasal polyps and marked septal deviation that significantly interfered with nasal air flow.
* in the opinion of the Investigator, were dependent upon nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* are on immunotherapy (desensitization therapy), unless on a regular maintenance schedule prior to the Screening visit and staying on this schedule for the remainder of the study. Subjects could not receive desensitization treatment within 24 hours prior to a study visit.
* smoke, or ex-smokers who had smoked within the previous six months.
* had current evidence of clinically significant hematopoietic, cardiovascular, hepatic, immunologic, renal, neurologic, psychiatric, autoimmune disease, or other disease that precludes the subject's participation in the study or with the subject's ability to complete the diary cards.
* were morbidly obese (BMI >= 35).
* were night-shift workers and those who did not have a standard asleep at night / awake during the day cycle.
* had any history of life threatening asthma attacks or subjects who had been treated in the emergency room or been admitted to the hospital for asthma control within the previous 3 months or more than once in the previous 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2003-07-01 (Actual); Primary Completion 2004-11-01 (Actual); Study Completion 2004-11-01 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 averaged over weeks 1 to 4. | Over weeks 1 to 4

SECONDARY OUTCOMES:
Change from Baseline in chest symptoms, nasal symptoms, and eye symptom scores | Day 15 and Day 29
Interference with sleep and daily activities | Day 15 and Day 29
Number of nocturnal awakenings due to chest symptoms | Day 15 and Day 29
Overall Therapeutic Response to therapy of allergic airway disease symptoms (investigator and joint evaluation) | Day 15 and Day 29
Change from Baseline in chest symptoms, nasal symptoms, and eye symptom scores | ALL TREATMENT VISITS (Day 1, Day 15, and Day 29)
Change in FEV1, FVC, FEF(25%-75%), PEFR | ALL TREATMENT VISITS (Day 1, Day 15, and Day 29)
Use of Proventil® HFA rescue medication | ALL TREATMENT VISITS (Day 1, Day 15, and Day 29)
Interference with sleep and daily activities | ALL TREATMENT VISITS (Day 1, Day 15, and Day 29)
Number of nocturnal awakenings due to chest symptoms | ALL TREATMENT VISITS (Day 1, Day 15, and Day 29)